CLINICAL TRIAL: NCT02461680
Title: Management Of The Partial Lesions Of The Fingers Flexor Tendons, Prospective Randomized Trial Of 2 Surgical Procedures: Tangential Resection Versus Direct Suture
Brief Title: Treatment for Partial Lesions of the Fingers Flexor Tendons : Tangential Resection or Direct Suture
Acronym: FLEXOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6021
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Flexor Tendon Injury; Lesions Of The Fingers Flexor Tendons
Keywords: partial section of the flexor tendons
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tangential resection (Experimental): the tendon's injury is treated with a tangential resection
  Interventions: Procedure: tangential resection
- Suture (Active Comparator): The tendon's injury is sutured
  Interventions: Procedure: suture

INTERVENTIONS:
Procedure: tangential resection — the tendon's injury is treated with a tangential resection performed with a surgical blade N°11 The shape of the tangential resection was adapted such that the cross-section disappered
  Arms: Tangential resection
Procedure: suture
  Arms: Suture

SUMMARY:
Flexors tendon injuries are frequent and serious with a potential of definitive functional aftereffects. In the case of partial injury, the treatment is debated. There are 2 techniques of possible repair, the direct suture and the tangential resection. The investigators have already demonstrated that this last technique was favorable for injuries going to 50 %. In the case of partial section between 50 and 75 %, the investigators think that the technique of tangential resection compared with the direct suture would not increase the risks of secondary breaks, would authorize even an immediate mobilization and would decrease the secondary complications.

The main objective is to highlight that the tangential resection is not lower than the classic technique on the clinical plan The secondary objectives are to highlight the non-inferiority of the tangential technique in clinical terms (pains, dexterity, complications), radiologics (MRI, ultrasound) and functional (function, go back to leisures and professional activities)

ELIGIBILITY:
Inclusion Criteria:

* wound dating less than 48 hours
* partial section from 50 % to 75 % of the flexor tendons (deep and/or superficial flexors, long flexor of the thumb) in zones 1, 2, 3, T1 and T2
* tendinous injuries on a single finger

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Total active motion Grasp | third month,
  Total active motion is the addition of angles in flexion of IPP, IPD and MCP joints of a finger in active mobility

CONTACTS AND LOCATIONS:
Overall Officials: Sybille FACCA, MD, Principal Investigator — CHU Strasbourg
Locations (1):
- CHU Strasbourg,, Strasbourg, France